CLINICAL TRIAL: NCT07105605
Title: The Effect of Peer Mentoring Program on Therapeutic Communication Skills of Students of Pediatric Nursing
Brief Title: The Effect of Peer Mentoring Program on Therapeutic Communication Skills of Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Rukiye Çelik, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025 - 846
Record Dates: First submitted 2025-06-03; First posted 2025-08-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Nurse-Patient Relations; Peer Mentoring; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: pediatric nursing student
Who Masked: Participant
Masking Description: 1. Intervention
  2. Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Control group
- Intervention Group (Experimental): Intervention Group
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — pediatric nursing student
  Arms: Intervention Group

SUMMARY:
The study was planned as a post-test randomized controlled experimental study with 70 students taking the Child Health and Diseases Nursing (CHN) course in the 2024-2025 academic year at Gazi University Faculty of Nursing. Before the CHN course, students were given the "Nursing The "Therapeutic Communication Skills Scale for Nursing Students" will be applied as a pre-test. Based on the scale scores, students will be assigned to intervention and control groups with simple randomization so that their group scores will be similar. Students in the control group will attend a theoretical lesson on topics such as inpatient child, age and period characteristics and communication with children within the scope of the ÇSHH course. Each student in this group will be evaluated in the scope of the clinical practice within the scope of the ÇSHH course and students will be asked to fill out the post-test of the "Therapeutic Communication Skills Scale for Nursing Students". Students in the intervention group will attend a theoretical lesson on topics such as inpatient child, age and period characteristics and communication with children within the scope of the ÇSHH course. After the lesson, the importance of TI, how it can be applied and sample materials will be conveyed to the students in the intervention group by their peers in one class hour. During the clinical practice process within the scope of the ÇSHH course to be held after the lesson, students in the intervention group will receive one-on-one AM from their peers at least 3 times. After the peer mentoring program is completed and the materials are developed, they will be asked to complete the final test of the "Therapeutic Communication Skills Scale for Nursing Students". In addition, the TI materials developed by the students in both groups will be independently evaluated by two pediatric nursing professors who are experts in their field, apart from the researchers, and the agreement between the two experts will be analyzed with the kappa test.

DETAILED DESCRIPTION:
There are differences in communication with children compared to adults. Communication with children; communication skills vary due to the communication methods they use, their ability to express themselves and age period characteristics. The nurse who cares for a child patient must have effective communication skills, especially techniques for providing comfortable communication, and therapeutic communication skills. Therapeutic communication, which has both data collection and therapeutic properties, is essential for optimal nursing care. Therapeutic communication (TI) is the constructive and supportive form of communication established by health professionals with the patient and their family. This communication aims to meet the emotional and psychological needs of individuals based on the foundations of empathy, trust, respect and understanding . Therefore, it is very important for nurses and nursing students to develop TI skills. Current literature emphasizes that the curriculum should be expanded with practices that improve the effective communication skills of nursing students . Although communication is an indispensable part of nursing, literature reports that adequate TI skills are lacking among nurses and nursing students . Students can be supported in TI with peer mentoring. Peer mentoring (PM) can effectively support student success in nursing education while promoting a culture of care and support. As a result of a study conducted with nursing students, it was found that AM has the capacity to reduce attrition rates and increase academic performance, as well as to create personal and professional qualities in first-year and upper-year nursing students. It is thought that this study will increase the quality of nursing education, improve students' TI skills, facilitate the use of the TI method in pediatric clinics, and enable students to communicate more effectively with children. The study was planned as a post-test randomized controlled experimental study with 70 students taking the Child Health and Diseases Nursing (CHN) course in the 2024-2025 academic year at Gazi University Faculty of Nursing. Before the CHN course, students were given the "Nursing The "Therapeutic Communication Skills Scale for Nursing Students" will be applied as a pre-test. Based on the scale scores, students will be assigned to intervention and control groups with simple randomization so that their group scores will be similar. Students in the control group will attend a theoretical lesson on topics such as inpatient child, age and period characteristics and communication with children within the scope of the ÇSHH course. Each student in this group will be evaluated in the scope of the clinical practice within the scope of the ÇSHH course and students will be asked to fill out the post-test of the "Therapeutic Communication Skills Scale for Nursing Students". Students in the intervention group will attend a theoretical lesson on topics such as inpatient child, age and period characteristics and communication with children within the scope of the ÇSHH course. After the lesson, the importance of TI, how it can be applied and sample materials will be conveyed to the students in the intervention group by their peers in one class hour. During the clinical practice process within the scope of the ÇSHH course to be held after the lesson, students in the intervention group will receive one-on-one AM from their peers at least 3 times. After the peer mentoring program is completed and the materials are developed, they will be asked to complete the final test of the "Therapeutic Communication Skills Scale for Nursing Students". In addition, the TI materials developed by the students in both groups will be independently evaluated by two pediatric nursing professors who are experts in their field, apart from the researchers, and the agreement between the two experts will be analyzed with the kappa test.

ELIGIBILITY:
Inclusion Criteria:

* Being a 3rd year nursing student,
* Having completed the self-awareness and communication course,
* Accepting the study,
* Completing the peer education program.

Exclusion Criteria:

* Not having attended the program or having dropped out halfway through,
* Having a GPA below 2,
* Being a repeat student,
* Having previously received training related to therapeutic communication.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Therapeutic Communication Skills Scale for Nursing Students | baseline, 3. month after the intervention
  Therapeutic Communication Skills Scale for Nursing Students, min:16 max:112, high score high skill
Therapeutic Communication Material Evaluation Checklist | 3. month after the intervention
  Therapeutic Communication Material Evaluation Checklist, min:0 max:100, high score high skill

CONTACTS AND LOCATIONS:
Overall Officials: Rukiye Çelik, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)